CLINICAL TRIAL: NCT05516732
Title: Evaluation of Serotonergic Neurotransmission in Premotor and Motor Parkinson's Disease.
Brief Title: Serotonin Release in Premotor and Motor PD
Acronym: FOX3
Status: Recruiting | Type: Observational
Sponsor: University of Exeter (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-21-16
Record Dates: First submitted 2022-08-24; First posted 2022-08-26 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Parkinson Disease; Parkinson's; Parkinson's Disease; Neurodegenerative Diseases; Neurodegeneration; Positron Emission Tomography
MeSH Terms: conditions — Parkinson Disease; Neurodegenerative Diseases; Nerve Degeneration | interventions — Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole; Spinal Puncture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Biosamples collected during this study will be blood, urine, and CSF. Blood biomarkers include routine clinical laboratory, DNA testing, and other analyses
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- SNCA (Alpha-synuclein gene): PET and SPECT molecular imaging and MRI; Clinical investigation and computerized neuropsychological testing; Collection of blood, urine and CSF biomarkers of PD pathology
  Interventions: Other: Positron Emission Tomography (PET) scan using CIMBI-36 tracer; Other: Magnetic Resonance Imaging (MRI) Scan; Other: Positron Emission Tomography (PET) scan using DASB tracer; Other: FP-CIT Single-photon Emission Computed Tomography (SPECT) scan; Other: Lumbar puncture
- Idiopathic Parkinson's Disease: PET and SPECT molecular imaging and MRI; Clinical investigation and computerized neuropsychological testing; Collection of blood, urine and CSF biomarkers of PD pathology
  Interventions: Other: Positron Emission Tomography (PET) scan using CIMBI-36 tracer; Other: Magnetic Resonance Imaging (MRI) Scan; Other: Positron Emission Tomography (PET) scan using DASB tracer; Other: FP-CIT Single-photon Emission Computed Tomography (SPECT) scan; Other: Lumbar puncture

INTERVENTIONS:
Other: Positron Emission Tomography (PET) scan using CIMBI-36 tracer — This scan creates images of regional serotonin release in by using a tracer compound called CIMBI to highlight the brains capacity to release serotonin.
Other: Magnetic Resonance Imaging (MRI) Scan — MRI (magnetic resonance imaging) uses magnets alongside radio waves to create pictures of the brain
Other: Positron Emission Tomography (PET) scan using DASB tracer — To create images of the brain using a tracer called DASB, which is a highly selective for serotonin transporters, this highlights serotonin terminals and neurons in the brain.
Other: FP-CIT Single-photon Emission Computed Tomography (SPECT) scan — A single-photon emission computerized tomography (SPECT) scan allows analysis of brain function by creating 3D Pictures using compounds called tracers.
Other: Lumbar puncture — A lumbar puncture invovles a thin needle is inserted between the bones in your lower spine using local anaesthetic. This allows the collection of Cerebrospinal fluid ( CSF)

SUMMARY:
In this study, the investigators aim to provide a deeper understanding of Parkinson's disease and find a biomarker of Parkinson's disease. This is done using imaging scans called Positron Emission tomography (PET), Single Photon Emission Computed Tomography (SPECT), and Magnetic Resonance Imaging (MRI). The findings will provide a deeper understanding of the brain changes in Parkinson's disease. More importantly, this study will help with the discovery and development of new medications aiming to delay progression of Parkinson's disease symptoms

DETAILED DESCRIPTION:
The purpose of this study is to find a biomarker for Parkinson's disease (PD). A biomarker is an indicator of the presence of a disease, that can be measured, and that is able to give information about the progression, or severity, of it.

The study visits will take place in London. There are three locations on Hammersmith hospital campus, that are located near to each other. The NIHR Imperial Clinical Research Facility and Invicro London for clinical and MRI and PET assessments, and Imperial Healthcare Nuclear Medicine Department for the SPECT scan.

Participants will attend 5 visits in a 3 month period. These visits include an initial consent and assessment visit where some blood samples will also be taken. The second visit involves a PET scan with the tracer DASB along with an MRI scan. The third visit involves two PET scans one in the morning, with CIMBI tracer, an injection of Dexamphetamine, and then a second with CIMBI tracer to make a comparison. The fourth visit involves a SPECT scan, and the fifth visit is optional and would be for a lumbar puncture visit. Each visit will last around 6 hours.

ELIGIBILITY:
Inclusion criteria-

* Subjects must understand the nature of the study and must provide signed and dated written HRA-approved informed consent in accordance with local regulations before any protocol-specific screening procedures are performed;
* Males and females, age 25-85 years, inclusive;
* Women of child-bearing potential must use protocol-defined contraceptive measures and must have a negative β-hCG test at screening. For sexually active subjects (except females of non-childbearing potential-e.g., at least 2 years postmenopausal or surgically sterile), condoms should be used in addition to other birth control methods for the duration of the study and for 3 months after the last administration of PET or SPECT ligands. These patients must be willing to remain on their current form of contraception for the duration of the study. All male subjects must agree to refrain from donating sperm for the duration of the study and for 3 months after the last administration of PET or SPECT ligands. Sexually active male subjects must agree to use condoms to protect their partners from becoming pregnant for the duration of the study and for 3 months after the last administration of PET or SPECT ligands (i.e. for 15 consecutive months following baseline PET and SPECT scans); agree to ensure that they and their partners are routinely using a medically approved contraceptive method. It is important that male subjects not impregnate others for the duration of the study and for 3 months after the last administration of PET or SPECT ligands;
* Able and willing to participate in all scheduled evaluations, abide by all study restrictions, and complete all required tests and procedures;
* Adequate visual and auditory acuity to complete the psychological testing;
* In the opinion of the investigator, the subject must be considered likely to comply with the study protocol and to have a high probability of completing the study.

Exclusion criteria -

* Subjects lacking capacity according to investigator judgement;
* Subjects taking serotonin acting drugs such as antidepressants (i.e. tricyclic or selective serotonin reuptake inhibitors etc.);
* Pregnancy or breastfeeding or intent to become pregnant in the next 18 months;
* Subjects with current or a recent history of drug or alcohol abuse/dependence;
* Subjects who have other neurological disorders and known intracranial co-morbidities such as stroke, hemorrhage, space-occupying lesions;
* Presence of any clinically significant medical condition (including cardiovascular, respiratory, cerebrovascular, hematological, hepatic, renal, gastrointestinal, or other disease) that, based on the judgment of the investigator, is clinically unstable, is likely to deteriorate during the course of the study, could put the patient at risk because of participation in the study, could affect the subject's ability to complete the study, or could influence the study results;
* History of suicidal behaviour or active suicidal ideation;
* Within 1 year prior to screen or between screen and baseline (Day -1), any of the following: myocardial infarction; hospitalization for congestive heart failure; hospitalization for, or symptoms of, unstable angina; or syncope not related to PD;
* History or presence of renal disease or impaired renal function;
* Clinically important infection (e.g., chronic, persistent, or acute infection) within 30 days prior to screen or between screen and baseline (Day -1);
* History of cancer within the last 5 years, with the exception of nonmetastatic basal cell carcinoma of the skin;
* Clinically significant blood clotting or bleeding disorder, including clinically significant abnormal findings in laboratory assessments of coagulation or hematology;
* Use of antipsychotic medication within 3 months prior to screen or between screen and baseline (Day -1);
* Use of any anticoagulant within 30 days prior to baseline and follow-up PET scans;
* Use of any oral corticosteroid within 30 days prior to baseline and follow-up PET scans;
* Use of metoclopramide within 30 days prior to baseline and follow-up (Day -1);
* Use of any thyroid medication within 30 days prior to baseline and follow-up (Day -1);
* Regular use (e.g., taken > 3 days/week) of narcotic pain medications within 30 days prior to baseline and follow-up (Day -1);
* Presence of any of the following MRI contraindications: pacemaker; cardiac defibrillator; spinal cord or vagus nerve stimulator; aneurysm clip; artificial heart valve; recent coronary or carotid stent; ear implant; CSF shunt; other implanted medical device (e.g., Swan-Ganz catheter, insulin pump); or metal fragments or foreign objects in the eyes, skin, or body;
* Negative modified Allen test in both hands, unless the brachial artery is used for arterial cannulation;
* Claustrophobia or history of back pain that makes prolonged laying on the PET or MRI scanner intolerable;
* History of severe skin allergy;
* Patients who had previous surgery for PD (including but not limited to deep brain stimulation [DBS] or cell transplantation);
* Patients who are treated with duodopa or apomorphine;
* Initiation or change in pharmacologic therapy for symptoms of PD within 30 days prior to screen or between screen and baseline and follow-up (Day -1).
* GDS score greater than or equal to 10 (GDS score of 5 - 9 requires Investigator discretion to enter study).
* STAI Form Y-1 greater than or equal to 54 requires Investigator discretion to enter study.

Ages: 25 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A cohort of carriers of genetic mutations for familial forms of Parkinson's Disease, Idiopathic Parkinson's Disease patients, and previously collected data from healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
DASB (a marker of Serotonin transporter) used to quantify in vivo pathology of serotonin | 3 Weeks
  To quantify serotonergic pathology with [11C]3-amino-4-(2- imethylaminomethylphenylsulfanyl)-benzonitrile (DASB) Positron Emission Tomography (PET)
SPECT to measure brain molecular pathology | 3 Weeks
  To quantify serotonergic pathology with [11C]DASB PET and dopaminergic pathology with Single-photon Emission Computed Tomography (SPECT)
Magnetic Resonance Imaging (MRI) | 3 Weeks
  Magnetic Resonance Imaging (MRI) to view structural and microstructural changes and structural connectivity.
CIMBI to measure serotonin release | 3 weeks
  CIMBI-36 can be interpreted to show serotonin release capacity both quantifiably and locational.

OTHER OUTCOMES:
Movement Disorder Society- Unified Parkinson's Disease Rating Scale (MDS-UPDRS) To determine if there is a correlation with neuropsychological and behavioural evaluation. | 3 Weeks
  A rating tool used to gauge the course of Parkinson's disease in patients
Montreal Cognitive Assessment (MOCA) to determine if there is a correlation with neuropsychological and behavioural evaluation | 3 Weeks
  A cognitive screening test designed to assist in the detection of mild cognitive impairment. Scored out of 30.
Cambridge Neuropsychological Test Automated Battery (CANTAB) to determine if there is a correlation with neuropsychological and behavioural evaluation | 3 Weeks
  Administered to detect cognitive issues & brain disorders efficiently.
Symbol Digit Modalities Test (SDMT) to determine if there is a correlation with neuropsychological and behavioural evaluation | 3 Weeks
  To be used in screening for organic cerebral dysfunction sored out of 110
Beck Depression Inventory-II (BDI-II) to determine if there is a correlation with neuropsychological and behavioural evaluation | 3 Weeks
  A brief, self-report inventory designed to measure the severity of depression symptomatology
State-Trait Anxiety Inventory (STAI) to determine if there is a correlation with neuropsychological and behavioural evaluation | 3 Weeks
  A commonly used measure of trait and state anxiety. Used to diagnose anxiety and to distinguish it from depressive syndromes.
University of Pennsylvania Smell Identification Test to determine if there is a correlation with neuropsychological and behavioural evaluation | 3 Weeks
  This is used to test the function of an individual's olfactory system
Movement Disorder Society- Non-Motor Symptoms scale for Parkinson's Disease MDS-NMSS to determine if there is a correlation with neuropsychological and behavioural evaluation | 3 Weeks
  This is a 30-item rater-based scale to assess a wide range of non-motor symptoms in patients with Parkinson's disease
Scales for Outcomes in Parkinson's Disease-Autonomic questionnaire - Autonomic Dysfunction (SCOPA-AUT) to determine if there is a correlation with neuropsychological and behavioural evaluation | 3 Weeks
  A 25 item assessment to evaluate autonomic symptoms in patients with Parkinson's disease

CONTACTS AND LOCATIONS:
Overall Officials: Marios M Politis, Professor, Principal Investigator — University of Exeter
Locations (1):
- University Of Exeter, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
to be decided

REFERENCES:
- See also: University of Exeter brief project information webpage — https://medicine.exeter.ac.uk/clinical-biomedical/research/nig/currentstudies/